CLINICAL TRIAL: NCT06461312
Title: Combined Pulsed Radiofrequency of the Pudendal Nerve With Ganglion Impar Block Effectively Alleviates Pudendal Neuralgia
Brief Title: Combined PRF of the Pudendal Nerve With Ganglion Impar Block Effectively Alleviates Pudendal Neuralgia
Acronym: PRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, director of department of Anesthesiology and Pain medicine, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB200-001
Record Dates: First submitted 2024-06-06; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Pudendal Neuralgia; Pulsed Radiofrequency
MeSH Terms: conditions — Pudendal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- enrolled patients (Experimental): Enrolled patients underwent pulsed radiofrequency of the pudendal nerve combined with ganglion impar block after pudendal nerve diagnostic block
  Interventions: Procedure: Combined pulsed radiofrequency of the pudendal nerve with ganglion impar block

INTERVENTIONS:
Procedure: Combined pulsed radiofrequency of the pudendal nerve with ganglion impar block — Combined pulsed radiofrequency of the pudendal nerve with ganglion impar block

SUMMARY:
Patients with pudendal neuralgia suffer from long-term pain, which severely affects their quality of life. Due to unclear etiology, there is a lack of specific treatment methods. The aim of this study is to evaluate the efficacy of combined pulsed radiofrequency with ganglion impar block therapy helps evaluate the effectiveness of this treatment method for pudendal neuralgia, comparing it with traditional treatments or single interventions, and providing guidance for clinical practice.

DETAILED DESCRIPTION:
We plan to enroll patients with pudendal neuralgia .Pre-treatment, we collected data including pain assessment, anxiety, depression, catastrophizing, and pain sensitivity scales. Treatment involved ultrasound-guided pudendal nerve pulsed radiofrequency and X-ray-guided ganglion impar block. The Patient Global Impression of Change (PGIC) and Numeric Rating Scale (NRS) were used as the main observation indicators to evaluate the treatment effect at 1, 2, 3, and 6 months postoperatively, followed by correlation analysis with the scores of relevant scales.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old;
2. Diagnosis of pudendal neuralgia meets the Nantes criteria. essential criteria include the following：1）Pain in the territory of the pudendal nerve；2） Pain is predominantly experienced while sitting；3) The pain does not wake the patient at night；4）Pain with no objective sensory impairment；5）Pain relieved by diagnostic pudendal nerve block；
3. Received conservative treatment for more than 3 months, and either had poor response to conservative treatment or intolerable medication side effects.
4. Capable of signing informed consent form.

Exclusion Criteria:

1. Pain caused by pelvic malignant diseases or autoimmune diseases;
2. Pain caused by pelvic surgery;
3. Taking anticoagulant drugs or having abnormal coagulation function;
4. Pregnancy;
5. Systemic infectious diseases;
6. Inability to complete scale assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Change | 1month
  0 -100%#0=no change,100%= complete relief of pain symptoms.
Patient Global Impression of Change | 2months
  0 -100%#0=no change,100%= complete relief of pain symptoms.
Patient Global Impression of Change | 3months
  0 -100%#0=no change,100%= complete relief of pain symptoms.
Patient Global Impression of Change | 6months
  0 -100%#0=no change,100%= complete relief of pain symptoms.

SECONDARY OUTCOMES:
Numeric Rating Scale | 1month
  0-10#0 =no pain, 10 = the most severe pain.
Numeric Rating Scale | 2months
  0-10#0 =no pain, 10 = the most severe pain.
Numeric Rating Scale | 3months
  0-10#0 =no pain, 10 = the most severe pain.
Numeric Rating Scale | 6months
  0-10#0 =no pain, 10 = the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Liu, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No